CLINICAL TRIAL: NCT04221282
Title: ZEBinix Retention Rate in Epilepsy in Elderly Patients
Brief Title: ZEBinix® Retention Rate in Epilepsy in Elderly Patients
Acronym: ZEBRE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Saint Joseph Saint Luc de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: ZEBRE
Record Dates: First submitted 2019-11-05; First posted 2020-01-09 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Epilepsy; Aging Disorder; Aging; Epilepsy; Seizure
Keywords: epilepsy; elderly; aging; zebinix; Eslicarbazepine acetate; tolerance; antiepileptic drug
MeSH Terms: conditions — Epilepsy | interventions — eslicarbazepine acetate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Epileptic elderly patients: Elderly patients with partial-onset seizures
  Interventions: Drug: Zebinix

INTERVENTIONS:
Drug: Zebinix — ESL will be initiated by the investigator in patients as a first line monotherapy or adjunctive therapy. ESL will be prescribed according to the usual care. Posology and method of administration of ESL are defined by the summary of product characteristics. Then, data on the efficacy of ESL will be collected.
  Other Names: Eslicarbazepine acetate (ESL)

SUMMARY:
The incidence of provoked and unprovoked seizures is known to increase with advancing age. Eslicarbazepine acetate (ESL) is one of the third generation of antiepileptic drugs (AEDs) that have been developed in the last ten years with a favorable safety profile. ESL is approved in Europe and the USA as adjunctive or monotherapy in adults with partial-onset seizures. Nevertheless, retrospective data in monotherapy condition in the elderly epileptic population are sparse. The aim of the ZEBRE study is to evaluate the efficacy and the safety of ESL in elderly epileptic patients (> 65 years). The completion of this study will provide crucial information on the most appropriate ESL treatment for elderly patients suffering from partial seizures.

DETAILED DESCRIPTION:
The ZEBRE (ZEBinix® Retention rate in epilepsy in Elderly patients) study is a prospective, multicenter, descriptive study. ESL will be prescribed according to the usual care. Posology and method of administration of ESL are defined by the summary of product characteristics.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 65 years
2. Ability of patient/legal representative to understand the study and to give his/her non-opposition (at the investigator's discretion)
3. Epilepsy with refractory partial-onset seizures with or without secondary generalization confirmed or with primary generalized tonic-clonic (PGTC) seizures
4. At least one seizure in the last three months
5. Treatment for partial-onset seizures with ESL as a first line monotherapy or with an adjunctive therapy

Exclusion Criteria:

1. History of ESL treatment
2. History of status epilepticus, seizures occurring in cluster, pseudo-seizures
3. History of severe hepatic impairment (aspartate aminotransferase (AST) and alanine aminotransferase (ALT) > 2 times ULN, gamma-glutamyltranspeptidase (GGT) > 5 times ULN)
4. History of severe renal impairment (clearance CLCR <30ml/min)
5. History of hypersensitivity to other carboxamide derivatives (e.g. carbamazepine, oxcarbazepine)
6. History of severe hyponatremia (< 120 mmol/L)
7. Second or third degree atrioventricular block
8. More than one other antiepileptic drug

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients ≥ 65 years that undergo at least one seizure in the last three months and with no history of ESL tratment or history of epilepsy status will be screened. ESL will be initiated by the investigator in patients with refractory partial seizures with or without generalized seizures or with PGTC seizures as a first line monotherapy or adjunctive therapy. In case of inefficacy or toxicity the dose of ESL will be gradually titrated up to 1 600 mg or titrated down to 600 mg, respectively.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Retention rate of ESL treatment as assessed by the number of patients that are still included in the study. | at the end of the study treatment, at 6 months
  The retention rate is representative of the effect of ESL since ESL will be pursued only if ESL has a sufficient efficacy without adverse effect. To evaluate the effect of ESL in elderly patients with partial-onset seizures, the retention rate will be measured after 6 months of treatment with ESL.

SECONDARY OUTCOMES:
Quality of life of patients as assessed by QOLIE-10 questionnaire | at each visits required by the study (baseline, 3 months and 6 months)
  QOLIE-10 (quality of life in epilepsy) is a quality of life questionnaire for adults with epilepsy. There are 10 questions about health and daily activities. All positive responses are lower numbers and all negative responses are higher numbers.
Quality of life of patients as assessed by QoL-AD questionnaire | at each visits required by the study (baseline, 3 months and 6 months)
  Some patients with epilepsy also have cognitive decline. QOL-AD (quality of life in Alzheimer'disease) measure quality of life in people with severe cognitive decline. A total score of 13-52, with higher scores indicating better QoL.
Quality of life of patients as assessed by NDDIE questionnaire | at each visits required by the study (baseline, 3 months and 6 months)
  NDDI-E (neurological disorder depression inventory for epilepsy) is used for detecting major depressive disorder; a total score above 15 should raise the suspicion of a major depressive episode.
Incidence of treatment- adverse events as assessed by adverse events reports | through study completion, an average of 6 months
  Number of patients with treatment-related adverse events will be reported to the pharmacovigilance department. Number of participants with abnormal laboratory values and/or adverse events that are related to treatment will be assessed.
Incidence of seizures as assessed by the occurrence of seizures | at each visits required by the study (baseline, 3 months and 6 months)
  The number and the type of seizures or the number of seizure free in elderly patients will be reported
Observance of the treatment as recorded by the control of the drug administration | through study completion, an average of 6 months
  The treatment delivery by the pharmacy be performed to assess the compliance of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Adrien DIDELOT, MD, PhD, Principal Investigator — Centre Hospitalier saint Joseph St Luc
Locations (1):
- Centre Hospitalier St Joseph St Luc, Lyon, France